CLINICAL TRIAL: NCT00188500
Title: Efficacy, Tolerability and Long-Term Adherence of a Modified Ketogenic Diet (Atkins) in the Management of Pharmacoresistant Epilepsy
Brief Title: Efficacy of Modified Ketogenic Diet (Atkins) in Management of Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-0027-AE
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-12-29 (Estimated); Status verified 2004-03

CONDITIONS: Epilepsy
Keywords: epilepsy; atkins diet
MeSH Terms: conditions — Epilepsy | interventions — Diet, High-Protein Low-Carbohydrate

INTERVENTIONS:
Behavioral: atkins diet
Behavioral: ability to follow low carbohydrate diet

SUMMARY:
The purpose of this study is to determine whether patients with uncontrolled epilepsy can follow a low carbohydrate diet long-term and if so, how will that diet affect their seizures

DETAILED DESCRIPTION:
In the management of drug-resistant epilepsy, many strategies have been examined. The Ketogenic Diet, high in fats and low in all other nutrients was observed to be of benefit. However, due to its complexedness and unpalatability, this diet is rarely used in the adult population. A recent small study showed seizure reduction with the Atkins Diet.

In this study, patients will be randomized into one of 2 groups- group 1 receiving limited dietary instruction for the Atkins Diet and group 2- receiving detailed dietary instruction. A seizure severity-matched control group will also take part. We will follow these patients over a period of 2 years looking at seizure frequency, weight, sustainability of the diet, effect on anti-epilepsy medication dosage, effect in cognition, quality of life and financial impact of the diet.

Patients will come to clinic to see the dietitian at specific intervals. cognitive testing will also be done at the beginning of the study and every 6 months thereafter. Patients will keep food charts, ketosis charts and seizure diaries.

ELIGIBILITY:
Inclusion Criteria:medically refractory partial epilepsy financial ability to pay for higher priced food

-

Exclusion Criteria:

* Low BMI

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-08; Study Completion 2005-09

PRIMARY OUTCOMES:
seizure reduction

SECONDARY OUTCOMES:
cognitive improvement

CONTACTS AND LOCATIONS:
Overall Officials: J Martin delCampo, Principal Investigator — UHN
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada